CLINICAL TRIAL: NCT02205372
Title: A Phase II, Randomised, Double-blind, Placebo-controlled Study of MT-3995 (Low Dose) in Subjects With Diabetic Nephropathy
Brief Title: Safety, Tolerability and Pharmacokinetic Study of MT-3995 at a Low Dose in Subjects With Diabetic Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-3995-J04
Record Dates: First submitted 2014-07-27; First posted 2014-07-31 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — apararenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MT-3995 (Experimental)
  Interventions: Drug: MT-3995
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-3995
  Arms: MT-3995
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and pharmacokinetics of MT-3995 in Subjects with Diabetic Nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 diabetes mellitus and diabetic nephropathy, who have been treated with a stable dose of angiotensin converting enzyme-inhibitor (ACE-I) or angiotensin II receptor blocker (ARB)
* Glycosylated haemoglobin (HbA1c) ≤10.5%
* Subject with albuminuria

Exclusion Criteria:

* Subjects with type 1 diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, secondary diabetes mellitus (Cushing's syndrome, steroidogenic diabetes).
* Serum potassium level <3.5 or >5.0 mmol/L
* Subjects who had acute kidney injury within 3 months prior to baseline or have undergone hemodialysis at any time prior to randomisation
* Subjects with clinically significant hypotension

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Frequency and nature of treatment-emergent adverse events and serious adverse events. | 20 weeks

SECONDARY OUTCOMES:
Plasma concentrations of MT-3995 | 20 weeks
Plasma concentrations of major metabolite of MT-3995 | 20 weeks
Change from baseline in Urine albumin-to-creatinine ratio (UACR) | 20 weeks
Change from baseline in blood pressure | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masaomi Nangaku, Professor, Study Director — Division of Nephrology and Endocrinology University of Tokyo School of medicine; Kazuoki Kondou, Adviｓer, Study Director — Tanabe Pharma Corporation
Locations (1):
- Touei Hospital, Sapporo, Hokkaido, Japan